CLINICAL TRIAL: NCT04235153
Title: CAncer, NUtrition and Taste - Validation of the CANUT-QVA Questionnaire on Eating Habits in Cancer Patients
Acronym: CANUT-QVA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0617
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Hematologic Cancer; Undernutrition; Chemotherapy Effect; Taste Disorders; Chemotherapy-Induced Change; Olfactory Disorder
MeSH Terms: conditions — Hematologic Neoplasms; Malnutrition; Taste Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with solid or hematological cancer: All the patients complete the CANUT-QVA questionnaire
  Interventions: Other: Evaluation of the 9 dimensions of the CANUT-QVA questionnaire

INTERVENTIONS:
Other: Evaluation of the 9 dimensions of the CANUT-QVA questionnaire — Evaluation of the contribution of a new questionnaire by patients with solid or hematological cancer according to 9 dimensions:
  1. Making food
  2. Place where the meals are eaten
  3. Eating and drinking: Nutrition
  4. Eating and drinking: The pleasure of tasting, chewing
  5. Eating and drinking: Satiated, well being
  6. Food preparation: Supply, choice, presentation
  7. Eating and drinking: Feelings
  8. After eating: heaviness, discomfort, hunger
  9. Taste/Odour Problems to confirm the number and structure of factors obtained at the end of the pre-study and to remove redundant questions.

SUMMARY:
Cancer patients are at high risk of undernutrition, which is generally more pronounced for solid tumours (upper digestive tract, Ear Nose and Throat (ENT), bronchial tubes). This undernutrition leads to major weight loss and cachexia, and may represent the first sign of a call for a diagnosis of cancer. Cancer-related undernutrition is multi-factorial origins and has multiple consequences.

Chemotherapy treatments can induce various adverse effects in patients, including sensory disturbances at the beginning of treatment in addition to disturbances that may already be present before any treatment. The alteration of taste and odour, observed in 86% of patients, can induce a change in food preferences, promote the development of aversions, and therefore, lead to a significant reduction in the pleasure of eating. Loss of appetite, decreased food intake and the development of aversions to certain foods are situations experienced by a large proportion of patients treated with chemotherapy.

The assessment of taste disorders in patients treated with chemotherapy is established through the use of questionnaires, interviews and taste tests.

Changes in the perception and identification of salty, sweet, bitter and sour flavours are common in patients treated with chemotherapy.

As regards food products, patients report developing olfactory hypersensitivity mainly for food of animal origin, in particular for odours of fish, frying, cheese and eggs.

The CANUT project aims to study the effect of pathology and chemotherapy on gustatory and olfactory mechanisms, and in particular on interindividual differences in the perception and appreciation of food.

In order to monitor the evolution of patients' eating habits over time, the diet-related quality of life questionnaire (CANUT-QVA) was constructed from items selected from the Well-being related to Food questionnaire (WELLBFQ) after eliminating questions that were too general or expressed in terms of importance to use perception-related responses as a priority.

After this part, an evaluation of the 9 dimensions of the CANUT-QVA questionnaire will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patient with solid or hematological cancer (any stage of disease and any treatment) diagnosed within 12 months of inclusion.
* Patient who does not object to participate in the trial
* Patient affiliated to a social security system

Exclusion Criteria:

* Minor patient (age <18 years).
* Patient under trusteeship, curatorship or protective measures.
* Patient who has already completed the questionnaire.
* Patient not sufficiently able to speak French to answer the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with solid or hematological cancer complete the CANUT-QVA questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Validate the 9 dimensions of the CANUT-QVA questionnaire identified during the general population analysis. | day 0
  The main evaluation criterion will be the adequacy between the responses to the food quality of life questionnaire by patients and the structure of the 9 dimensions as presented in the context (relevance of the questions for each dimension).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Groupement Hospitalier Lyon Sud, Service pneumologie, Pierre-Bénite, France